CLINICAL TRIAL: NCT04443608
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Phase 4 Study of the Efficacy & Safety of Patiromer for Oral Suspension in Combination With Standard of Care Treatment in ED Patients With Hyperkalemia
Brief Title: Patiromer Utility as an Adjunct Treatment in Patients Needing Urgent Hyperkalemia Management
Acronym: PLATINUM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment window ended
Sponsor: Comprehensive Research Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRA-US-001
Record Dates: First submitted 2020-06-08; First posted 2020-06-23 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-04

CONDITIONS: Hyperkalemia
Keywords: potassium; dialysis; emergency department
MeSH Terms: conditions — Hyperkalemia; Emergencies | interventions — Suspensions; patiromer; Bulk Drugs

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Veltassa (Active Comparator): 3 packets of study drug powder will be mixed with a liquid (water, apple or cranberry juice) and given to patient to drink while in the emergency department
  Interventions: Drug: Patiromer Powder for Oral Suspension [Veltassa]
- Placebo (Placebo Comparator): 3 packets of study drug powder will be mixed with a liquid (water, apple or cranberry juice) and given to patient to drink while in the emergency department
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Patiromer Powder for Oral Suspension [Veltassa] — Powder will be mixed with a liquid (water, apple or cranberry juice) and given to patient to drink
  Other Names: Active drug
  Arms: Veltassa
Drug: Placebo — Powder will be mixed with a liquid (water, apple or cranberry juice) and given to patient to drink
  Other Names: Inactive substance
  Arms: Placebo

SUMMARY:
When a patient arrives to an emergency department and is found to have an elevated potassium level in the blood, there is no one standardized treatment, therefore it is not known if one treatment is superior to other. The purpose of this study is to help determine if a drug called patiromer (already approved by the FDA) can help lower potassium levels while patients are in the emergency department.

DETAILED DESCRIPTION:
Given the lack of consistency in hyperkalemia treatment in the ED and the high cost of emergent dialysis, there is a need for the development and systematic evaluation of a treatment protocol to shift potassium into the cells followed by the removal of potassium from the body with a potassium binder.. The present study will use a systematic approach to shifting potassium into the cells followed by binding potassium in the gastrointestinal tract in hyperkalemic patients presenting to the ED. Study subjects will receive patiromer or placebo to determine if patiromer reduces the need for additional medical intervention for the management of hyperkalemia in patients initially treated with IV and inhaled therapy in the ED.

Upon enrollment, patiromer will be administered at a dose selected because of its safety and efficacy shown in a pilot study named REDUCE.

Up to 300 patients will be enrolled and followed for up to 14 days, and potassium levels will be measured at pre-determined intervals to assess drug's impact. concomitant medications will be recorded to help determine if study drug helped, not just lower hyperkalemia, but also decrease the number of total interventions needed to reach a normal potassium level.

ELIGIBILITY:
Inclusion Criteria:

* Hyperkalemia, defined as K+ ≥5.8 obtained via local laboratory or point-of-care testing
* Written informed consent obtained.

Exclusion Criteria:

1. Clinically significant arrhythmia, defined as any arrhythmia requiring ongoing IV antiarrhythmic therapy.
2. Patients who are hemodynamically unstable, defined as mean arterial pressure ≤65 mmHg or heart rate ≤40 beats per minute or ≥125 beats per minute at time of screening
3. Hyperkalemia solely due to overdose on potassium supplements
4. Known bowel obstruction
5. Subjects currently being treated with or having taken potassium binders (e.g., patiromer, sodium or calcium polystyrene sulfonate or sodium zirconium cyclosilicate) in the 7 days prior to baseline
6. Subjects expected to receive dialysis during the first 6 hours of the study treatment period
7. Known hypersensitivity to patiromer or its ingredients
8. Participation in any other investigational device or drug study <30 days prior to screening, or current treatment with other investigational agent(s)
9. Inability to consume the investigational product or, in the opinion of the Investigator unsuitable for study participation
10. Life expectancy of less than 6 months
11. Patients with automatically timed medication orders to control potassium in the ED
12. Patient is known to be pregnant or breastfeeding
13. An employee of investigational site or sponsors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
The need for additional potassium-lowering medical interventions | Duration of patient's emergency department visit, up to 6 hours
  Net clinical benefit (mean difference in number of interventions less change in serum potassium)

SECONDARY OUTCOMES:
Potassium level trends after receiving study drug | Up to 24 hours after study drug dose is given
  Proportion of subjects without post-baseline potassium-related medical interventions at Hours 4, 6 and 8
Potassium level trends after receiving study drug | 4 hours
  Net clinical benefit at Hour 4
Potassium level trends after receiving study drug | ED visit, up to 10 hours
  Number of post-baseline potassium-related medical interventions up until Hours 4, 6, and 8 and ED discharge
Potassium level trends after receiving study drug | 8 hours
  Proportion of subjects with sustained potassium reduction (defined as K+ ≤5.5 mEq/l and 4 hours without potassium-related medical intervention) at Hours 6 and 8
Potassium level trends after receiving study drug | Up to 24 hours after study drug dose is given
  K+ 24 hours after ED discharge

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Stanford University School of Medicine, Stanford, California
  - Yale University, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - George Washington University, Washington D.C., District of Columbia
  - Baystate Medical Center, Springfield, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University of St Louis, St Louis, Missouri
  - Mt Sinai. Icahn School of Medicine, New York, New York
  - Maimonides Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University. Wexner Medical Center, Columbus, Ohio
  - JPS Health Network, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rafique Z, Budden J, Quinn CM, Duanmu Y, Safdar B, Bischof JJ, Driver BE, Herzog CA, Weir MR, Singer AJ, Boone S, Soto-Ruiz KM, Peacock WF. Patiromer utility as an adjunct treatment in patients needing urgent hyperkalaemia management (PLATINUM): design of a multicentre, randomised, double-blind, placebo-controlled, parallel-group study. BMJ Open. 2023 Jun 12;13(6):e071311. doi: 10.1136/bmjopen-2022-071311. PMID 37308268